CLINICAL TRIAL: NCT04698902
Title: Influence of Calcium Pattern on Plaque Modification Achieved With Intracoronary Lithotripsy
Status: Completed | Type: Observational
Sponsor: Fundacion Investigacion Interhospitalaria Cardiovascular (Other)
Responsible Party: Principal Investigator, Nieves Gonzalo, Dr., Fundacion Investigacion Interhospitalaria Cardiovascular
Other Study IDs: 20/599-E
Record Dates: First submitted 2021-01-05; First posted 2021-01-07 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Coronary Artery Disease; Intracoronary Lithotripsy; Optical Coherence Tomography; Percutaneous Coronary Intervention; Calcification; Stent
MeSH Terms: conditions — Coronary Artery Disease; Calcinosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Circumferential calcification: Patients with circumferential pattern of coronary artery calcification by OCT (Optical coherence tomography) assessment (arc of calcium >180 degrees)
  Interventions: Device: Intracoronary lithotripsy
- Eccentric calcification: Patients with an eccentric pattern of coronary artery calcification by OCT (Optical coherence tomography) assessment (arc of calcium <180 degrees)
  Interventions: Device: Intracoronary lithotripsy
- Nodular calcification: Patients with calcium nodules identified by OCT (Optical coherence tomography) assessment
  Interventions: Device: Intracoronary lithotripsy

INTERVENTIONS:
Device: Intracoronary lithotripsy — Intracoronary lithotripsy involves the use of sonic pressure waves generated from emitters enclosed within a balloon delivery system. The generated sonic waves act to fracture calcium within the coronary artery wall.

SUMMARY:
Calcified coronary artery disease is a frequently encountered problem that can lead to poorer outcomes for patients undergoing PCI. Recently, intravascular lithotripsy has become available for the treatment of callcified coronary artery disease. The effect of intravascular lithotripsy on varying calcium patterns has not been adequately explored.

This is an investigator initiated, open label, non-blinded, observational study involving a number of centers in Spain examining the effect of intravasuclar lithotripsy in varying calcium patterns. 100 patients wll be enrolled. Optical coherence tomography will be used to assess the effect of intravascular lithotripsy on varying calcium patterns (concentric, eccentric and nodular).

DETAILED DESCRIPTION:
Calcified coronary artery disease continues to present a challenge for Interventional Cardiologists. Moderate calcification is found in over 25% of coronary artery lesions planned for percutaneous coronary intervention (PCI). Outcomes for patients undergoing PCI to calcified lesions have been shown to be consistently poorer than in non-calcified lesions. Recently, intravascular lithotripsy has become available for the treatment of calcified coronary artery disease. The effect of intravascular lithotripsy on varying calcium patterns has not been adequately explored.

This is an investigator initiated, open label, non-blinded, observational study involving a number of centers in Spain. Patients with an indication of PCI and with a significant calcium burden requiring modification will be invited to participate. PCI procedures will be performed via either radial or femoral access as deemed appropriate by the operator and in accordance with local protocols. Intravascular imaging using OCT will be performed prior to calcium modification to define the pattern of calcium, after calcium modification to assess the effectiveness of IVL therapy and after stent implantation to assess stent expansion.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years of age
* Patients with an indication for PCI (ischemic symptoms or evidence of myocardial ischemia (inducible or spontaneous) in the presence of >50% de novo severely calcified coronary stenosis that requires IVL treatment.

Exclusion Criteria:

* Patients unwilling or unable to sign informed consent for the procedure
* Patients with severe peripheral vascular disease limiting vascular access to the extent that it is unsafe to perform the procedure
* Patients with severe renal dysfunction (eGFR <15mls/min and not receiving dialysis)
* Treatment of vessels < 2.5mm diameter which are not amenable to IVL treatment or OCT assessment.
* Treatment of lesions located very distally in the coronary vessel where the OCT catheter may not reach.
* Inability to cross the lesion with the OCT catheter due to very severe stenosis or severe vessel tortuosity.
* Ostial left main stem or right coronary artery lesions which may be difficult to visualise by OCT
* Patients requiring concomitant use of rotational or orbital atherectomy of LASER.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with calcified coronary artery disease planned for percutaneous coronary intervention and stenting with the use of intravascular lithotripsy for calcium modification prior to stenting.
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Percentage of lesions with Calcium Fractures | At the time of percutaneous coronary intervention
  Percentage of lesions showing calcium modification (fractures) after intravascular lithotripsy (IVL) in nodular eccentric and concentric calcium patterns

SECONDARY OUTCOMES:
Number of calcium fractures | At the time of percutaneous coronary intervention
  Number of calcium fractures visible on OCT after IVL treatment
Number of quadrants with calcium fractures | At the time of percutaneous coronary intervention
  Number of quadrants with calcium fractures after IVL treatment as assessed by OCT
Calcium modification in eccentric versus concentric calcium | At the time of percutaneous coronary intervention
  Percentage of lesions with calcium arc <180 versus >180 degrees with fractures as assessed by OCT
Stent expansion | At the time of percutaneous coronary intervention
  Percentage stent expansion in patients with and without calcium modification (fractures) after application of IVL
Stent symmetry | At the time of percutaneous coronary intervention
  Stent symmetry index in patients with and without calcium modification (fractures) after IVL application
Stent symmetry | At the time of percutaneous coronary intervention
  Stent symmetry index in patients with concentric versus eccentric calcification

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clínico San Carlos, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided